CLINICAL TRIAL: NCT06319105
Title: Accelerating the Path To Scale for Injectable PrEP in Malawi: An Implementation Evaluation
Brief Title: PathToScale: An Implementation Evaluation
Status: Recruiting | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: AIDS Vaccine Advocacy Coalition (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency); Center for the Development of People (Unknown); Cooper/Smith (Unknown); Elizabeth Glaser Pediatric AIDS Foundation (Other); Family Health Services (Unknown); Healthqual (Unknown); Johns Hopkins Research Project, Malawi (Unknown); Johns Hopkins Bloomberg School of Public Health (Other); Kamuzu University of Health Sciences (Other); Blantyre District Health Office, Malawi (Unknown); Lilongwe District Health Office, Malawi (Unknown); Lighthouse Trust (Other); Ministry of Health, Malawi (Other Government); National AIDS Commission, Malawi (Unknown); Pakachere Institute of Health and Development Communication (Unknown); Partners in Hope, Inc. (Industry); Population Services International (Other); University of North Carolina (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); United States President's Emergency Plan for AIDS Relief (U.S. Federal Agency); Quantitative Engineering Design (Unknown); Clinton Health Access Initiative-Malawi (Unknown)
Responsible Party: Principal Investigator, Charles Holmes, Director, Center for Innovation in Global Health, Georgetown University
Other Study IDs: 775736
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Oral Pre-exposure Prophylaxis (PrEP); Long-acting Injectable Cabotegravir for PrEP
Keywords: HIV; pre-exposure prophylaxis (PrEP); Implementation Science; Long-acting injectable cabotegravir for PrEP; Oral pre-exposure prophylaxis (PrEP)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Standard intervention: Offer PrEP choice: Offer pre-exposure prophylaxis choice between oral and long-acting injectable cabotegravir for pre-exposure prophylaxis across 36 study sites.
  Interventions: Other: Standard intervention: Offer PrEP choice

INTERVENTIONS:
Other: Standard intervention: Offer PrEP choice — This hybrid observational-implementation study will observe the implementation of a choice of oral pre-exposure prophylaxis or long-acting injectable cabotegravir for pre-exposure prophylaxis for all participants.

SUMMARY:
The purpose of this study is to evaluate the implementation and clinical outcomes of expanded pre-exposure prophylaxis delivery modalities and service delivery points offering long-acting injectable cabotegravir and oral pre-exposure prophylaxis to high-priority groups through diverse delivery channels.

DETAILED DESCRIPTION:
This study will assess client uptake, equitable reach, and continuation of oral and injectable pre-exposure prophylaxis implementation across priority populations and service delivery channels in real-world settings. The study will also evaluate long-acting injectable cabotegravir for pre-exposure prophylaxis implementation readiness and implementation outcomes across these delivery channels and priority populations from the perspectives of providers and clients. Demand generation activities will also be evaluated. Lastly, the study will conduct clinical surveillance of long-acting injectable cabotegravir outcomes at scale, including pregnancy outcomes among clients who become pregnant or are pregnant on long-acting injectable cabotegravir, and seroconversion and resistance outcomes of long-acting injectable cabotegravir users.

This study takes a hybrid observational-implementation approach, which will leverage routine programmatic data from pre-exposure prophylaxis implementation from national registries and tools from the real-world roll-out of long-acting injectable cabotegravir and will complement these routine data with targeted collection of implementation outcomes and barriers and facilitators to implementation with a subset of stakeholders. Research staff will not implement long-acting injectable cabotegravir, but rather long-acting injectable cabotegravir will be implemented by the Ministry of Health and implementing partners under routine care and following the Ministry of Health pre-exposure prophylaxis guidelines.

Per the Ministry of Health eligibility guidelines, we anticipate the following populations will be prioritized for long-acting injectable cabotegravir for pre-exposure prophylaxis distribution nationally, following individual risk assessment.

* Female sex workers (FSW)
* Men who have sex with men (MSM)
* Transgender individuals (TG)
* Women and adolescent girls and young women (AGYW) presenting at sexually transmitted infection (STI) services
* Breastfeeding women
* Male partners of female sex workers (FSW)
* Men at high risk, presenting with a syndromic or lab-confirmed sexually transmitted infection (STI)

Pre-exposure prophylaxis users will be passively enrolled into the evaluation. Routine, de-identified programmatic data will be utilized from Ministry of Health pre-exposure prophylaxis ScanForms to identify the number and demographic characteristics (gender, age, indication for pre-exposure prophylaxis) of oral and long-acting injectable cabotegravir for pre-exposure prophylaxis users initiating pre-exposure prophylaxis modalities by site, switching from oral to long-acting injectable cabotegravir for pre-exposure prophylaxis (and vice versa), and continuation rates.

Additional data collection activities will be conducted to evaluate the process of implementation and its fidelity, including facility context assessments, a long-acting injectable cabotegravir for pre-exposure prophylaxis provision readiness assessment with providers across implementing facilities, qualitative interviews with providers, observational assessments of providers across facilities, and client exit interviews.

Primary Outcomes

Outcome 1 Title: Pre-exposure prophylaxis uptake by modality Description: Comparison of pre-exposure prophylaxis uptake by modality (injectable vs. oral) between months 7-12 Timeframe: 12 months after enrollment Analysis: Pre-exposure prophylaxis uptake across modalities will be described overall as the average proportion taking up injectable vs. oral pre-exposure prophylaxis per site, and compared across sites using proportion-tests.

Outcome 2 Title: Pre-exposure prophylaxis uptake by delivery channel Description: Comparison of oral and injectable pre-exposure prophylaxis uptake by service delivery channel (e.g. HIV counseling and testing, postnatal care, family planning, sexually transmitted infection clinics, drop-in centers, youth-friendly services, etc.) Timeframe: 12 months after enrollment Analysis: Monthly counts of pre-exposure prophylaxis uptake by delivery channel will be described and compared using Poisson regression adjusting for HIV testing service eligible-site volume and available supply; clustering within sites will be included.

Outcome 3 Title: Pre-exposure prophylaxis uptake by population Description: Comparison of oral and injectable pre-exposure prophylaxis uptake by pre-exposure prophylaxis client population (e.g. female sex workers, breastfeeding women, adolescent girls and young women/women at high risk for HIV infection, men who have sex with men, transgender persons, men at high risk for HIV acquisition).

Timeframe: 12 months after enrollment Analysis: Monthly counts of pre-exposure prophylaxis uptake by population will be described and compared using Poisson regression adjusting for HIV testing service eligible-site volume and available supply; clustering within sites will be included.

Outcome 4 Title: Pre-exposure prophylaxis continuation by modality Description: Comparison of pre-exposure prophylaxis continuation by modality (injectable vs. oral) Timeframe: 12 months after enrollment Analysis: Proportion of clients persisting on pre-exposure prophylaxis across each time point will be described and compared by modality using log-binomial regression adjusting for number of pre-exposure prophylaxis clients at the site by modality; clustering within sites will be included.

Outcome 5 Title: Pre-exposure prophylaxis continuation by delivery channel Description: Comparison of pre-exposure prophylaxis continuation by channel (e.g. HIV counseling and testing, post-natal care, family planning, sexually transmitted infection clinics, drop-in centers, youth-friendly services, etc.) Timeframe: 12 months after enrollment Analysis: Proportion of clients persisting on pre-exposure prophylaxis across each time point will be described and compared by delivery channel using log-binomial regression adjusting for number of pre-exposure prophylaxis clients at the site by modality; clustering within sites will be included.

Outcome 6 Title: Pre-exposure prophylaxis continuation by population Description: Comparison of pre-exposure prophylaxis continuation by pre-exposure prophylaxis client population (e.g. female sex workers, breastfeeding women, adolescent girls and young women/women at high risk for HIV acquisition, men who have sex with men, transgender persons, men at high risk for HIV acquisition).

Timeframe: 12 months after enrollment Analysis: Proportion of clients persisting on pre-exposure prophylaxis across each time point will be described and compared by population using log-binomial regression adjusting for number of pre-exposure prophylaxis clients at the site by modality; clustering within sites will be included.

Outcome 7 Title: Rates of switching between oral and injectable pre-exposure prophylaxis Description: Describe rates of switching between oral and injectable pre-exposure prophylaxis among pre-exposure prophylaxis users Timeframe: 18 months after enrollment Analysis: Describe overall switching proportion to oral and injectable pre-exposure prophylaxis at 18-months and compare proportions of those switching using proportions testing clustered on site

Secondary Outcomes Outcome 8 Title: Implementation readiness Description: Implementation readiness across sites and service delivery channels using Normalisation MeAsurement Development questionnaire (NoMAD) scores Timeframe: 6 months after enrollment Analysis: Describe mean implementation readiness scores across sites and compare across service delivery channels using analysis of variance (ANOVA) testing.

Outcome 9 Title: Pregnancy rates among long-acting injectable cabotegravir for pre-exposure prophylaxis users Description: Incidence of pregnancy among long-acting injectable cabotegravir for pre-exposure prophylaxis users Timeframe: 18 months after enrollment Analysis: Describe pregnancies per 100-woman years of follow-up among cisgender women on long-acting injectable cabotegravir

Outcome 10 Title: Pregnancy outcomes among long-acting injectable cabotegravir for pre-exposure prophylaxis users Description: Describe birth registry outcomes among long-acting injectable cabotegravir for pre-exposure prophylaxis users Timeframe: 18 months after enrollment Analysis: Proportion of pregnancy abnormalities will be described overall amongst cisgender women with incident long-acting injectable cabotegravir pregnancies and compared to women with oral pre-exposure prophylaxis pregnancies using comparison of proportions.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for long-acting injectable cabotegravir for pre-exposure prophylaxis will be applied per Ministry of Health guidelines. Per Ministry of Health guidelines, the following populations will be prioritized for long-acting injectable cabotegravir for pre-exposure prophylaxis distribution, following individual risk assessment:

Individuals who are 15+ years old AND either

1. Female sex workers (FSW) OR
2. Men who have sex with men (MSM) OR
3. Transgender individuals (TG) OR
4. Women and adolescent girls and young women (AGYW) presenting at STI services and/or family planning and/or HIV testing services OR
5. Breastfeeding women (BFW) OR
6. Male partners of female sex workers and/or Men at high risk for HIV and/or men presenting with a syndromic or lab-confirmed sexually transmitted infections. All individuals initiated on long-acting injectable cabotegravir for pre-exposure prophylaxis 15 years or above will be included in the passively enrolled sample.

Exclusion Criteria:

* Per Ministry of Health guidelines, exclusion criteria for long-acting injectable cabotegravir for pre-exposure prophylaxis includes:

Those living with HIV-1 or evidence of possible acute HIV infection OR Those with a prior Hepatitis B diagnosis OR Those with a known history of severe side effects to Cabotegravir Long Acting OR Those unwilling or unable to return for 3-monthly HIV testing or 2-monthly counseling and safety monitoring visits OR Clients currently on multi-drug resistance tuberculosis (MDR-TB) medications OR Clients currently taking post-exposure prophylaxis.

Ages: 15 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Active participants will be pre-exposure prophylaxis providers and clients from the 36 implementation facilities and key stakeholders (e.g. governmental and non-governmental stakeholders), who are invited to participate in study activities about their perspectives, prescribing and use of pre-exposure prophylaxis across the 36 PathToScale sites.
Sampling Method: Non-Probability Sample
Enrollment: 9900 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Pre-exposure prophylaxis uptake by modality | 12 months after enrollment
  Comparison of pre-exposure prophylaxis uptake by modality (injectable vs. oral) between months 7-12
Pre-exposure prophylaxis uptake by delivery channel | 12 months after enrollment
  Comparison of oral and injectable pre-exposure prophylaxis uptake by service delivery channel (e.g. HIV counseling and testing, postnatal care, family planning, sexually transmitted infection clinics, drop-in centers, youth-friendly services, etc.)
Pre-exposure prophylaxis uptake by population | 12 months after enrollment
  Comparison of oral and injectable pre-exposure prophylaxis uptake by pre-exposure prophylaxis client population (e.g. female sex workers, breastfeeding women, adolescent girls and young women/women at high risk for HIV infection, men who have sex with men, transgender persons, men at high risk for HIV acquisition).
Pre-exposure prophylaxis continuation by modality | 12 months after enrollment
  Comparison of pre-exposure prophylaxis continuation by modality (injectable vs. oral)
Pre-exposure prophylaxis continuation by delivery channel | 12 months after enrollment
  Comparison of pre-exposure prophylaxis continuation by channel (e.g. HIV counseling and testing, post-natal care, family planning, sexually transmitted infection clinics, drop-in centers, youth-friendly services, etc.)
Pre-exposure prophylaxis continuation by population | 12 months after enrollment
  Comparison of pre-exposure prophylaxis continuation by pre-exposure prophylaxis client population (e.g. female sex workers, breastfeeding women, adolescent girls and young women/women at high risk for HIV acquisition, men who have sex with men, transgender persons, men at high risk for HIV acquisition).
Rates of switching between oral and injectable pre-exposure prophylaxis | 18 months after enrollment
  Describe rates of switching between oral and injectable pre-exposure prophylaxis among pre-exposure prophylaxis users

SECONDARY OUTCOMES:
Implementation readiness | 6 months after enrollment
  Implementation readiness across sites and service delivery channels using Normalisation MeAsurement Development questionnaire (NoMAD) scores
Pregnancy rates among long-acting injectable cabotegravir for pre-exposure prophylaxis users | 18 months after enrollment
  Incidence of pregnancy among long-acting injectable cabotegravir for pre-exposure prophylaxis users
Pregnancy outcomes among long-acting injectable cabotegravir for pre-exposure prophylaxis users | 18 months after enrollment
  Describe birth registry outcomes among long-acting injectable cabotegravir for pre-exposure prophylaxis users

CONTACTS AND LOCATIONS:
Overall Officials: Charles Holmes, MD, MPH, Principal Investigator — Georgetown University
Locations (1):
- Community Health Science Unit, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. We are working with vulnerable populations and can make aggregate data available by request. Approval from principal investigators will be necessary to release de-identified data.